CLINICAL TRIAL: NCT01066533
Title: Histologic and Immunohistochemical Study of Fibronectin and Tenascin in Human Teeth Pulp Capped With MTA and NEC
Brief Title: Immunohistochemical Study of Human Teeth Pulp Capped With Mineral Trioxide Aggregate (MTA) and Novel Endodontic Cement (NEC)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: immunohistochemistry markers are not recieved yet
Sponsor: Mashhad University of Medical Sciences (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Bahareh Joshan, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 583
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2009-07

CONDITIONS: Direct Pulp Capping
Keywords: MTA; NEC; Immunohistochemistry; fibronectin; tenascin

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mineral Trioxide Aggregate(MTA) (Experimental): MTA is a proper material for direct pulp capping,treatment of tooth perforations,root end filling.It is a safe and biocompatible material,which can induce cementum formation on root surface.In direct pulp capping, MTA can induce dentinal bridge formation on the expose surface to preserve pulp vitality.Although MTA has superior biocompatibility compared with the conventional materials,it has a delayed setting time, poor handling characteristics and off-white color
  Interventions: Other: direct pulp capping and covering the exposed pulp
- NEC cement (Experimental): NEC cement is a proper material for direct pulp capping and treatment of tooth perforation. It is a new dental material that combines reasonable biocompatibility of MTA with appropriate setting time,handling characteristics,chemical properties and color.Like MTA, NEC cement can induce dentinal bridge formation in direct pulp capping to preserve pulp vitality.
  Interventions: Other: direct pulp capping and covering the exposed pulp

INTERVENTIONS:
Other: direct pulp capping and covering the exposed pulp — In this arm 16 premolar teeth scheduled for extraction for orthodontic reasons were used.After signed consent was given by patients,local anesthesia was applied before operative procedures. Operative procedures were performed with rubber dam placement and disinfected with 2% chlorhexidine gluconate. Class I occlusal cavities were prepared with ¼ round carbide burs under air-distilled water cooling. At the exposure site hemorrhage was controlled by sterile cotton pellets, saline and 5.25% NaOCl.In this group MTA was mixed on a slab according to manufacture's instructions.Then MTA was carried with a carrier to exposed pulp and it was packed with a slight pressure by moist cotton pellet to completely cover the exposed pulp.The cavities were sealed immediately with Fuji II glass ionomer.The teeth were then followed and extracted(8 teeth after 2 weeks and 8 teeth after 8 weeks)
  Arms: Mineral Trioxide Aggregate(MTA)
Other: direct pulp capping and covering the exposed pulp — In this arm 16 premolar teeth scheduled for extraction for orthodontic reasons were used.All the procedure was carried the same as the other group.But NEC cement was used as pulp capping material.It was mixed with its liquid to provide a dense creamy mixture and then was applied on exposed pulp.the cavities were immediately sealed with Fuji II glass ionomer.The patients were followed and 8 teeth were extracted after 2 weeks and 8 teeth were extracted after 8 weeks.
  Arms: NEC cement

SUMMARY:
The purpose of this study is to evaluate the response of human dental pulp to capping with MTA and NEC by histology and immunohistochemistry, using fibronectin and tenascin as markers, following 2 weeks and 8 weeks.

DETAILED DESCRIPTION:
Capping of the exposed pulp is indicated for reversible pulp tissue injury after physical or mechanical trauma in developing or mature teeth.The response to direct pulp capping with materials such as MTA or NEC is the formation of dentin barrier, resulting from the recruitment and proliferation of undifferentiated cells.

Different materials can be used to induce dentinal bridge formation.MTA has been introduced as a proper material to induce dentinal bridge formation,with greater mean thickness of dentinal bridge and less inflammation compared to traditional materials like calcium hydroxide. Although biocompatible, MTA has a poor handling characteristic, delay setting time, off-white color, and it is almost expensive.The Novel Endodontic Cement (NEC) has been introduced to combine reasonable characteristics of MTA with appropriate chemical properties, setting time, color, and handling characteristics.

The extracellular matrix (ECM) of pulp comprises a variety of proteins and polysaccharides, forming a neat network. The ECM components can induce either reactionary or reparative dentin formation. Fibronectin (FN) and tenascin (TNC) are the two major glycoproteins involved in wound healing and odontogenesis.

Fibronectins (FNs) are a class of high molecular weight adhesive proteins composed of two very large subunits. It has a variety of cell functions, such as adhesion, migration, growth, and differentiation. Furthermore FN may be involved in the polarization and migration of odontoblasts.

Tenascin is a large oligomeric glycoprotein of the ECM secreted by fibroblasts and glial cells in tissue cultures. It has also been identified in pulp and more prominent in dentinogenesis. TN has been shown to be important in the differentiation of odontoblasts. Therefore, it may be associated with secondary dentin formation, when pulp cells differentiate into odontoblasts in response to physiologic stimuli.

Although dentin bridge formation has been reported,using different materials such as MTA and NEC in direct pulp cap, but the exact mechanism is not well understood. Immunohistochemistry, using different markers, may be useful in developing the molecules involved in this process.

Moreover,response of dental pulp to different pulp capping materials can be studied,including mean thickness of dentinal bridge, morphology of dentinal bridge, and intensity of pulp inflammation and presence of odontoblast cells.

ELIGIBILITY:
Inclusion Criteria:

* patients 16-30 year-old
* patients with no systemic disease
* vital mature teeth with closed apex, no caries either clinically or radiographically, and without any restoration
* patients willing to participate in study

Exclusion Criteria:

* patients not in the range of 16-30 year-old
* patients with systemic disease
* nonvital teeth
* open apex teeth
* teeth with caries or restorations
* patients not willing to participate in study

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
histologic study of: 1-mean thickness of formed dentinal bridge 2-morphology of formed dentinal bridge 3-intensity of pulp inflammation 4-odontoblastic layer | 2 weeks and 8 weeks

SECONDARY OUTCOMES:
expression of Fibronectin and Tenascin by immunohistochemistry on a scale of 1 to 3: (a) 1 equals no staining; (b) 2 equals light-medium staining; (c) 3 equals medium-heavy staining for the marker | 2 weeks and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Javidi, endodontist, Study Director — Mashhad University of Medical Sciences; Mohamad hasan zarrabi, endodontist, Study Director — Mashhad University of Medical Sciences
Locations (1):
- Mashhad university of medical sciences, Mashhad, Khorasan, Iran